CLINICAL TRIAL: NCT04039932
Title: Faith Leaders Advocating for Maternal Empowerment (FLAME)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Gondar (Other)
Responsible Party: Principal Investigator, Brandon Guthrie, Assistant Professor, School of Public Health, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001662
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Prenatal Care; Maternal Health Services; Perinatal Care

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial assigning facility catchment areas to intervention vs. standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: FLAME
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: FLAME — The FLAME intervention trains pairs of faith leaders and community health workers and deploys them to conduct behavior change outreach in their communities.
  Arms: Intervention

SUMMARY:
In 2015, the average Ethiopian woman had a 1 in 64 lifetime risk of death due to complications of childbirth and 87,414 newborns died before their 28th day of life. Demand for MNCH services, however, remains low in Ethiopia's rural communities most at risk with only 16% of women delivering in a health facility.

The investigator's project responds to the challenge of creating demand for existing MNCH services in rural Ethiopia, which fell short of reaching Millennium Development Goal targets for reducing preventable maternal and neonatal deaths. This study addresses two strategic drivers to prevent maternal mortality identified by USAID including improving individual, household, and community behaviors and norms and increasing equity of access and use of services by the most vulnerable.

The primary objective of the study is to determine the impact of a behavior change intervention that partners Ethiopian Orthodox priests with members of the Health Development Army (HDA) and trains them to conduct maternal health outreach to increase births attended by skilled health personnel among women who attend ≥1 ANC visits.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Willing to receive intervention counseling

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Limited to pregnant women with female sex assigned at birth
Enrollment: 18 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Facility delivery | Through study completion, an average of 18 months
  The proportion of births attended by skilled health personnel among the women who attended ≥1 ANC visits

SECONDARY OUTCOMES:
Any ANC | Through study completion, an average of 18 months
  Number of women who attended ≥1 ANC visits
Complete ANC | Through study completion, an average of 18 months
  Number of women who attended ANC 4

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Guthrie, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Gondar, Gonder, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guthrie BL, Tsegaye AT, Rankin KC, Walson JL, Alemie GA. Partnering faith leaders with community health workers increases utilization of antenatal care and facility delivery services in Ethiopia: A cluster randomized trial. J Glob Health. 2021 Oct 30;11:04063. doi: 10.7189/jogh.11.04063. eCollection 2021. PMID 34737863